CLINICAL TRIAL: NCT04250558
Title: Indocyanine Green Fluorescence Guided Imaging in Lower Extremity Amputation Patients
Brief Title: ICG Fluorescence Imaging in Lower Extremity Amputation Patients
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Staff Physician, Dartmouth-Hitchcock Medical Center
Other Study IDs: D20046
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Trauma Injury
Keywords: Trauma; Amputation; Orthopaedic; Lower Extremity
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Lower Extremity Amputation — patients 18 years of age or older who will have a planned lower leg (either below knee, through knee, or above knee) amputation surgery are scheduled to undergo a lower extremity amputation (either below knee, through knee or above knee), performed by a participating surgeon or delegate. Provision of informed consent.

SUMMARY:
This is a non-randomized prospective study of 30 patients scheduled to undergo lower extremity amputation (below the knee, through the knee or above the knee) evaluating bone perfusion and viability using indocyanine green (ICG) fluorescence imaging at several steps during surgical procedure.

DETAILED DESCRIPTION:
This is a non-randomized prospective study of 30 patients scheduled to undergo lower extremity amputation (below the knee, through the knee or above the knee) evaluating bone perfusion and viability using indocyanine green (ICG) fluorescence imaging at several steps during surgical procedure. The data collected in this study will inform the development of methodology and thresholds around providing surgeons with objective data regarding critically injured bone in the setting of musculoskeletal trauma and/or bone infection. This will improve our management of and decrease variation associated with management of these disabling conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Scheduled for a lower extremity amputation (either below knee, through knee or above knee)
3. Provision of informed consent

Exclusion Criteria:

1. Iodine allergy
2. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients 18 years of age or older who present to DHMC and are scheduled to undergo a lower extremity amputation (either below knee, through knee or above knee) will be considered for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Extremity Amputation: Patients over 18 undergoing lower extremity amputation
Period: Overall Study
Arm/Group | Extremity Amputation
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Extremity Amputation: Patients over 18 undergoing either below knee, through knee, or above knee lower extremity amputation.
Arm/Group | Extremity Amputation
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Total Bone Blood Flow [Median (Full Range); unit: mL/min/100g] — measured as mL/min/100g
  mL/min/100g | 6.7 [0 to 30]

OUTCOME MEASURES:

1. Primary Outcome: Total Bone Blood Flow (TBBF)-Post Osteotomy
Description: Changes to total bone blood flow changes that occur as a result of osteotomy and soft tissue stripping associated with the amputationas will be assessed by immunofluorescence based dynamic constrast enhanced fluorescence imaging.
Time Frame: 4 hours
Measure: Median (Full Range); unit: mL/min/100g
Arm/Group | Extremity Amputation
Number analyzed (Participants) | 15
mL/min/100g | 4.9 [0 to 30]

2. Primary Outcome: Total Bone Blood Flow (TBBF)-Post Osteotomy+Stripping
Description: Changes to total bone blood flow changes that occur as a result of osteotomy and soft tissue stripping associated with the amputations will be assessed by immunofluorescence based dynamic contrast enhanced fluorescence imaging.
Time Frame: 4 hours
Measure: Median (Full Range); unit: mL/min/100g
Arm/Group | Extremity Amputation
Number analyzed (Participants) | 15
mL/min/100g | 0.8 [0 to 30]
Statistical Analysis 1: Comparison: Extremity Amputation; Kinetic parameters were assessed by Mann-Whitney U test in MATLAB Statistics and Machine Learning Toolbox. Receiver operating characteristic (ROC) analysis based on logistic regression was utilized, with one surgical condition versus the other two states as the binary dependent variable, and each perfusion-related kinetic parameter of Imax, IS and BF as the independent variable. Power analysis was performed to evaluate the statistical validity, using G*Power software; Test type: Other; p = 0.05, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 0-30 minutes post infusion
Description: Per clinicaltrials.gov defintions
Arm/Group | Extremity Amputation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04250558/Prot_000.pdf